CLINICAL TRIAL: NCT03836937
Title: Role of Obeticholic Acid in the Patients of NAFLD With Raised ALT- A Randomized Clinical Control Trial Study
Brief Title: Role of Obeticholic Acid in the Patients of NAFLD With Raised ALT
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Salimullah Medical College Mitford Hospital (Other Government)
Responsible Party: Principal Investigator, Md. Fazal Karim, Associate Professor, Sir Salimullah Medical College Mitford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirSalimullahMCMH
Record Dates: First submitted 2019-01-09; First posted 2019-02-11 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid

STUDY DESIGN:
Intervention Model Description: Open label randomized clinical control trial study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obeticholic acid (Experimental): Patients diagnosed as NAFLD with raised ALT will be treated with both life style modification and Obeticholic acid. Obeticholic acid will be given as 10 mg twice daily. Life style modification includes moderate exercise that is 30 minutes brisk walking a day with dietary advice to avoid fatty foods and excessive sugar containing diet and intake of at least 3 vegetables per day.
  Interventions: Drug: Obeticholic acid
- Lifestyle modification (No Intervention): Patients diagnosed as NAFLD with raised ALT will be given only life style modification.Life style modification includes moderate exercise that is 30 minutes brisk walking a day with dietary advice to avoid fatty foods and excessive sugar containing diet and intake of at least 3 vegetables per day.

INTERVENTIONS:
Drug: Obeticholic acid — Farnesoid X receptor ligand which is a semi synthetic bile acid analogue
  Other Names: Life style modification
  Arms: Obeticholic acid

SUMMARY:
This study will be conducted upon the patients with fatty liver disease. Patients who will be diagnosed as a case of fatty liver disease by ultrasound with raised liver enzyme (ALT) will be primarily selected for the study. A total number of 70 patients will be randomly selected for the study that will also be divided into two groups for the study purpose. The patients will be informed about the details of the study. After getting the detail information those who will give informed written consent will be finally included in the study. One group of patients will be treated by both life style modification and Obeticholic acid. Another group of patients by only life style modification. After 3 months of treatment the two groups will be compared of improvement of fatty liver disease and liver enzyme by improvement of fibroscan with CAP value as well as improvement of ALT value.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an increasingly common cause of chronic liver disease worldwide and it is associated with increased liver-related mortality and hepatocellular carcinoma, even in the absence of cirrhosis. The prevalence of NAFLD is steadily increasing and is currently 20%-30% in Western countries and 5%-18% in Asia. It progresses to cirrhosis in 15-20% of affected individuals and is a rising indication for liver transplantation. NAFLD is the commonest cause of elevated liver enzymes. Lifestyle modifications, including diet and exercise, are imperative for achieving weight loss and reducing insulin resistance and hepatic steatosis and inflammation in patients with NAFLD. But are suboptimal by long-term adherence in patients with NAFLD. On the other hand, current pharmacological treatment of NAFLD has limited efficacy and unfavorable safety profile. In this context, obeticholic acid, a selective agonist of the farnesoid X receptors, might represent a useful option in these patients. Preclinical studies suggest that obeticholic acid improves hepatic steatosis, inflammation and fibrosis. A randomized, placebo-controlled Farnesoid X Receptor Ligand Obeticholic Acid in non-alcoholic steatohepatitis Treatment (FLINT) trial also showed improvements in liver histology in patients with NAFLD who received obeticholic acid. So, there is a need to develop more effective and safe agents for this common and life-threatening disease.

Farnesoid X receptor (FXR) is a member of the nuclear receptor super family expressed in the liver, kidney, intestine and adrenal glands. In addition to regulation of bile acid (BA) synthesis, several lines of evidence have suggested that FXR plays a role in the pathophysiology of NAFLD/NASH. Obeticholic acid is a synthetically modified bile acid that is a potent agonist of the farnesoid X nuclear receptor (FXR), a nuclear receptor with major effects on bile acid synthesis and transport as well as lipid metabolism and glucose homeostasis. Obeticholic acid has been shown to improve serum enzymes in several diseases including nonalcoholic fatty liver disease and primary biliary cirrhosis. In FLINT trial treatment with obeticholic acid (25 mg/day for 72 weeks) resulted in a highly statistically significant improvement in the NAFLD Activity Score of at least two points, with no worsening of fibrosis. 45% (50 of 110) of the treated group had this improvement compared with 21% (23 of 109) of the placebo-treated controls.

The objective of the study will be to assess the efficacy of obeticholic acid on improvement of NAFLD and ALT values in patients with fatty liver disease.

The study will be conducted in the department of Hepatology, Sir Salimullah Medical College and Mitford Hospital. It will be a randomized open label clinical control trial study. Patients diagnosed with non-alcoholic fatty liver disease (NAFLD) will be initially targeted for the study. Patients who will be diagnosed as a case of NAFLD by ultrasound with raised Alanin aminotransferase (ALT) (>40 U/L) will be primarily selected for the study. The total sample size will be 70 that will be divided into two groups (Group-A and Group-B) for the study purpose. The patients will be informed about the details of the study. After getting the detail information, those who will give informed written consent will be finally included in the study. A series of baseline investigations including CBC with ESR, fasting blood sugar (FBS), 2 hours after 75 g glucose, alanine aminotransferase (ALT), aspartate-aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), bilirubin (B), PT with INR, serum albumin, total cholesterol (TC) & triglycerides (TG), LDL-C, HDL-C, Thyroid function test will be determined on fresh serum using an auto-analyzer. Fibroscan with CAP as well as ALT will be done to assess the baseline status of the patients at the time of enrollment of the study. Group-A patients will be treated by both life style modification and Obeticholic acid and Group-B patients by only life style modification. We shall give 10 mg obeticholic acid twice daily to the patients of Group-1. Life style modification including moderate exercise that is 30 minutes brisk walking a day with dietary advice to avoid fatty foods and excessive sugar containing diet and intake of at least 3 vegetables per day will be advised to all the patients in both Groups. The patients will be followed for 3 months. Patients will come for follow-up after 1 month and finally after 3 months. Each visit will take place between 10.00 am to 02.00 p.m. & consist with a clinical examination, blood pressure (BP) & body mass index (BMI) determinations and a questionnaire. BMI will be computed using the formula: [weight (kg)]/ [square of height (meters)]. Serum will be collected for CBC with ESR, FBS, 2 hours after 75 g glucose, ALT, AST, PT with INR, serum albumin, GGT, TC, TG, HDL, LDL in first and last visit. An alcohol consumption questionnaire will also be administered in each visit and study compliance will be strictly monitored. After 3 months of treatment the two groups will be compared of improvement of NAFLD and liver enzyme by improvement of fibroscan with CAP value as well as improvement of ALT value with the baseline ALT and fibroscan with CAP values.

All Data will be presented as mean ± SD & analyzed by SPSS (version 23). Qualitative data will be analyzed by Chi-square test & quantitative data will be analyzed by student's t-test. A statistically significant result will be considered when P value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD (by USG)
* Raised ALT (>40 U/L)

Exclusion Criteria:

* Patient with significant alcohol intake (more than 20 gm/day).
* Patient with history of taking drugs that may cause fatty liver (i.e. tamoxifen, valproic acid, amiodarone, methotrexate, steroid, OCP) or history of taking drugs that have shown benefit in previous NASH pilot studies (i.e. vitamin E, metformin, thiazolidinediones, statin, ARB, fibrates, DPP-4 inhibitor, Omega-3 fatty acid).
* Chronic viral hepatitis (HBV, HCV).
* Pregnancy
* Patient with co-morbid condition (COPD, CKD, CCF etc.)
* Patient with history of recent MI
* Patient with liver failure
* Patient with hypothyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fibroscan score (Kpa) and CAP value (Kpa) which signifies fibrosis and steatosis status respectively. | For 12 weeks from the date of enrollment of the patient.
  Obeticholic acid and life style modification improve fibroscan with CAP results in patients with NAFLD.
  1. Change in symptoms after 12 weeks of treatment or life style modification.
  2. Change in liver function test, fibroscan values and CAP values after treatment or life style modification.
Change in BMI (weight in kg/height in meter square) | For 12 weeks from the date of enrollment of the patient.
Change in ALT (U/L) | For 12 weeks from the date of enrollment of the patient.
Fasting blood sugar (FBS) (mmol/L) | For 12 weeks from the date of enrollment of the patient.
2 hours after 75 gm glucose (mmol/L) | For 12 weeks from the date of enrollment of the patient
Serum bilirubin (mg/dl) | For 12 weeks from the date of enrollment of the patient
Aspertate aminotransferase (AST) (U/L) | For 12 weeks from the date of enrollment of the patient
Gamma glutamyle transpeptidase (GGT) (U/L) | For 12 weeks from the date of enrollment of the patient
Serum albumin (gm/dl) | For 12 weeks from the date of enrollment of the patient
Prothrombin time (PT) (sec) | For 12 weeks from the date of enrollment of the patient
Total cholesterol (mg/dl) | For 12 weeks from the date of enrollment of the patient
Triglyceride (TG) (mg/dl) | For 12 weeks from the date of enrollment of the patient
LDL cholesterol (mg/dl) | For 12 weeks from the date of enrollment of the patient
HDL cholesterol (mg/dl) | For 12 weeks from the date of enrollment of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Md F Karim, MBBS,FCPS,MD, Principal Investigator — Sir Salimullah Medical College
Locations (1):
- Department of Hepatology, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study and statistical analysis, the study report will be published
Supporting Information: CSR
Time Frame: February'2019-June'2019
Access Criteria: drfazalkarim@gmail.com

REFERENCES:
- [Background] Neuschwander-Tetri BA, Loomba R, Sanyal AJ, Lavine JE, Van Natta ML, Abdelmalek MF, Chalasani N, Dasarathy S, Diehl AM, Hameed B, Kowdley KV, McCullough A, Terrault N, Clark JM, Tonascia J, Brunt EM, Kleiner DE, Doo E; NASH Clinical Research Network. Farnesoid X nuclear receptor ligand obeticholic acid for non-cirrhotic, non-alcoholic steatohepatitis (FLINT): a multicentre, randomised, placebo-controlled trial. Lancet. 2015 Mar 14;385(9972):956-65. doi: 10.1016/S0140-6736(14)61933-4. Epub 2014 Nov 7. PMID 25468160
- [Background] Makri E, Cholongitas E, Tziomalos K. Emerging role of obeticholic acid in the management of nonalcoholic fatty liver disease. World J Gastroenterol. 2016 Nov 7;22(41):9039-9043. doi: 10.3748/wjg.v22.i41.9039. PMID 27895393
- [Background] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166
- [Background] Kirk E, Reeds DN, Finck BN, Mayurranjan SM, Patterson BW, Klein S. Dietary fat and carbohydrates differentially alter insulin sensitivity during caloric restriction. Gastroenterology. 2009 May;136(5):1552-60. doi: 10.1053/j.gastro.2009.01.048. Epub 2009 Jan 25. PMID 19208352